CLINICAL TRIAL: NCT02866942
Title: Safety of Nasal Influenza Immunisation in Children With Asthma - The SNIFFLE-4 Study
Brief Title: Safety of Nasal Influenza Immunisation in Children With Asthma
Acronym: SNIFFLE-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Principal Investigator, Paul Turner, MRC Clinician Scientist, Imperial College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16SM3348; 2016-002352-24 (EudraCT Number)
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Asthma (Experimental): LAIV administration in children with asthma receiving treatment according to British Thoracic Society step 2+
  Interventions: Drug: Administration of Live attenuated influenza vaccine (LAIV)

INTERVENTIONS:
Drug: Administration of Live attenuated influenza vaccine (LAIV)
  Other Names: Flumist; Fluenz

SUMMARY:
A new influenza vaccine, known as LAIV (Live Attenuated Intranasal Vaccine) has recently been approved by a number of licensing boards and is given by a spray into the nose. In the United Kingdom (UK), the vaccine has been demonstrated to be highly effective against influenza infection. Further, despite concerns that LAIV can cause wheezing in children under age 2 years, the previous SNIFFLE studies have demonstrated it to be safe in children over 2 years with mild-moderate asthma.

The objective of this multicentre study is to further assess the safety of intranasal LAIV in children with asthma and recurrent wheeze, including those with severe symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 - 18 years old (inclusive)
* Physician diagnosis of asthma or recurrent wheezing (by the hospital specialist) AND (i) in children age 2-4 years: ≥2 exacerbations in the past year requiring oral steroids or observation in-hospital beyond 4 hours duration, OR (ii) in children ≥ 5 years of age, receiving treatment equivalent to at least BTS/SIGN step 2 therapy.
* Written informed consent from parent/guardian (or the patient themselves from age 16 years), with assent from children aged 8 years and above wherever possible.

Exclusion Criteria:

1. Admission to Paediatric Intensive Care for invasive ventilation due to a respiratory illness in the preceding 2 years.
2. Contraindications to LAIV (notwithstanding allergy to egg protein), which include:

   1. Hypersensitivity to the active ingredients, gelatin or gentamicin (a possible trace residue)
   2. Previous systemic allergic reaction to LAIV
   3. Previous allergic reaction to an influenza vaccine (not LAIV) is a relative contra-indication, which must be discussed with the site PI to confirm patient suitability
   4. Children/adolescents who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and high-dose corticosteroids**.

      **High-dose steroids is defined as a treatment course for at least one month, equivalent to a dose greater than 20mg prednisolone per day (any age), or for children under 20kg, a dose greater than 1mg/kg/day.

      NB: LAIV is not contraindicated for use in individuals with asymptomatic HIV infection; or individuals who are receiving topical/inhaled/low-dose oral systemic corticosteroids or those receiving corticosteroids as replacement therapy, e.g. for adrenal insufficiency.
   5. Children and adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wild-type influenza infection.
   6. pregnancy
3. Contraindications to vaccination on that occasion, e.g. due to child being acutely unwell:

   1. Febrile ≥38.0 degrees C in last 72 hours
   2. *Acute wheeze in last 72 hours requiring treatment beyond that normally prescribed for regular use by the child's treating healthcare professional
   3. *Recent admission to hospital in last 2 weeks for acute asthma
   4. *Current oral steroid for asthma exacerbation or course completed within last 2 weeks
   5. Any other significant condition or circumstance which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

      * Items 3b-3d are relative contra-indications: Many children with "difficult-to-control" symptoms may meet fail to meet these criteria on a routine basis. Where these are present, the study centre PIs are able to authorise participation on a case-by-case basis, after assessing the child and their lung function at the time of enrolment.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 479 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, Principal Investigator — Imperial College London / Imperial College Healthcare NHS Trust / Public Health England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turner PJ, Southern J, Andrews NJ, Miller E, Erlewyn-Lajeunesse M; SNIFFLE Study Investigators. Safety of live attenuated influenza vaccine in atopic children with egg allergy. J Allergy Clin Immunol. 2015 Aug;136(2):376-81. doi: 10.1016/j.jaci.2014.12.1925. Epub 2015 Feb 13. PMID 25684279
- [Background] Turner PJ, Southern J, Andrews NJ, Miller E, Erlewyn-Lajeunesse M; SNIFFLE-2 Study Investigators. Safety of live attenuated influenza vaccine in young people with egg allergy: multicentre prospective cohort study. BMJ. 2015 Dec 8;351:h6291. doi: 10.1136/bmj.h6291. PMID 26645895
- [Derived] Jackson D, Pitcher M, Hudson C, Andrews N, Southern J, Ellis J, Hoschler K, Pebody R, Turner PJ, Miller E, Zambon M. Viral Shedding in Recipients of Live Attenuated Influenza Vaccine in the 2016-2017 and 2017-2018 Influenza Seasons in the United Kingdom. Clin Infect Dis. 2020 Jun 10;70(12):2505-2513. doi: 10.1093/cid/ciz719. PMID 31642899

RESULTS

PARTICIPANT FLOW:
Groups:
- Asthma: LAIV administration in children with asthma receiving treatment according to British Thoracic Society step 2+
  Administration of Live attenuated influenza vaccine (LAIV)
Period: Overall Study
Arm/Group | Asthma
Started | 479
Completed | 478
Not Completed | 1
Not completed — Invalid consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Asthma
Number analyzed (Participants) | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 476
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 9.3 [2.0 to 18.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 288
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 478
British Thoracic Society (BTS) Treatment Step 4+ [Count of Participants; unit: Participants] — STEP 4+, assigned as "persistent poor control" in asthma, is defined as:
  * requiring high dose inhaled corticosteroids (>800 micrograms beclomethasone equivalent) per day, and/or
  * 3+ preventer medications
  Participants | 229

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Symptoms and Control Pre and 4 Weeks Post LAIV, as Assessed by Validated Questionnaire
Description: The validated questionnaire to be used will depend on the age of the enrolled child:
  * Age 2-4 years: TRACK questionnaire
  * Age 5-11 years: Children's Asthma Control Test (C-ACT) score
  * Age 12+ years: Asthma Control Test (ACT) score
  The change in score (using the appropriate questionnaire for age) between pre- and 4 weeks post LAIV will be used to assess the primary outcome across all participants. a change in (c-)ACT of at least 3 points, or 10 points for TRACK will be determined a significant change.
  For TRACK, the minimum and maximum score possible is 0 and 100 respectively, the higher the score, the better is symptom control.
  For c-ACT, the minimum and maximum score possible is 0 and 27 respectively, the higher the score, the better controlled are asthma symptoms.
  For ACT, the minimum and maximum score possible is 5 and 25 respectively, the higher the score, the better controlled are asthma symptoms.
Time Frame: 4 weeks post LAIV
Population: 4 week follow-up data available in 319/478 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma
Number analyzed (Participants) | 319
Participants
  Improvement >= MID | 28
  No change | 254
  Deterioration >= MID | 37
Statistical Analysis 1: Comparison: Asthma; Test type: Other; p = 0.26, McNemar

2. Secondary Outcome: Incidence of Adverse Events (AE) and Serious Adverse Events (SAEs) in Children Receiving LAIV
Description: Incidence of a 'significant exacerbation' in asthma, defined as:
  i. At least 3 day course of oral steroids following an unscheduled contact with a healthcare professional; OR ii. Unscheduled visit to an Emergency department or admission to hospital for treatment of asthma symptoms, requiring systemic corticosteroids
Time Frame: Up to 4 weeks post LAIV administration
Measure: Count of Participants; unit: Participants
Arm/Group | Asthma
Number analyzed (Participants) | 319
Participants | 47

ADVERSE EVENTS:
Time Frame: 72 hours post LAIV administration
Arm/Group | Asthma
All-Cause Mortality (participants affected / at risk) | 0/478
Serious Adverse Events (participants affected / at risk) | 4/478
Other Adverse Events (participants affected / at risk) | 150/478
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asthma (N=478)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asthma (N=478)
Malaise (General disorders) | 42 (42)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 54 (54)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (27)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT02866942/Prot_SAP_000.pdf